CLINICAL TRIAL: NCT02770677
Title: Modified Dantien Salee Yoga Training Program in Chronic Obstructive Pulmonary Disease Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Duangjun Phantayuth, Assistant Professor, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MU-CIRB 2015/133.2808
Record Dates: First submitted 2016-04-20; First posted 2016-05-12 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Yoga; COPD; rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Detail of intervention is Yoga training program. 3 times /week ,12 weeks .
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Control group will be asked to continue their normal daily life without Yoga training
- Yoga group (Experimental): Yoga group will be exposed to Modified Dantien Salee Yoga Training Program for 12 weeks
  Interventions: Other: Modified Dantien Salee Yoga Training Program

INTERVENTIONS:
Other: Modified Dantien Salee Yoga Training Program — The intervention aims to improve pulmonary function and functional fitness.
  Arms: Yoga group

SUMMARY:
COPD patients will be recruited and assigned into one of each group: 1) Control group or 2) Yoga group. In Yoga groups, subjected will be asked to participate in Modified Dantien Yoga training for 12 weeks (3 times/week, 60 min/time). The subjects will be evaluated their pulmonary function, functional fitness performance, dyspnea score, and quality of life at baseline and after 12 wk training.

ELIGIBILITY:
Inclusion Criteria:

1. Stable COPD patients > or equal 6 weeks.
2. Age > or equal 50-80 years.
3. FEV1 > or equal 30% predicted after take bronchodilators drug.
4. Resting SpO2 > or equal 90% room air.
5. Did not pulmonary rehabilitation program before start the yoga

Exclusion Criteria:

1. Subjects with musculoskeletal disorders, mental and neurological disorders, and acute coronary heart disease.
2. Blood Pressure (systolic) > 180 mmHg.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-04-07 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline FVC (Forced Vital Capacity) (L) at 12 weeks | 12 weeks
  Change of FVC (Forced Vital Capacity) will be measured on a computerized Spirometer at the baseline and 12 weeks.
Change from baseline FEV1 (Forced Expiratory Volume in 1 minute)(L) at 12 weeks | 12 weeks
  Change of Forced Expiratory Volume in 1 second will be measured on a computerized Spirometer at the baseline and 12 weeks.
Change from baseline TLC (Total Lung Capacity) (L) at 12 weeks | 12 weeks
  Change of TLC (Total Lung Capacity) (L) will be measured on a computerized Spirometer at the baseline and 12 weeks.
Change from baseline FRC (Functional Residual Capacity) (L) at 12 weeks | 12 weeks
  Change of FRC (Functional Residual Capacity) (L) will be measured on a computerized Spirometer at the baseline and 12 weeks.
Change from baseline IC (Inspiratoy Capacity) (L) at 12 weeks | 12 weeks
  Change of IC (Inspiratoy Capacity) (L) will be measured on a computerized Spirometer at the baseline and 12 weeks.
Change from baseline RV (Residual Volume) (L) at 12 weeks | 12 weeks
  Change of RV (Residual Volume) (L) will be measured on a computerized Spirometer at the baseline and 12 weeks.
Change from baseline MVV (Maximum Voluntary Ventilation) (L/min) at 12 weeks | 12 weeks
  Change of MVV (Maximum Voluntary Ventilation) (L/min) will be measured on a computerized Spirometer at the baseline and 12 weeks.
Change from baseline PEFR (Peak Expiratory Flow Rate) (L/sec) at 12 weeks | 12 weeks
  Change of MVV (Maximum Voluntary Ventilation) (L/sec) will be measured on a computerized Spirometer at the baseline and 12 weeks.
Change from baseline DLCO (Diffusion capacity to carbon monoxide) (ml/mmHg/min) at 12 weeks | 12 weeks
  Change of DLCO (Diffusion capacity to carbon monoxide) (ml/mmHg/min) will be measured on a computerized Spirometer at the baseline and 12 weeks.
Change from baseline PI max (Maximal Inspiratoy Pressure) (cm H2O) at 12 weeks | 12 weeks
  Change of PI max (Maximal Inspiratoy Pressure) (cm H2O) will be measured on a computerized Spirometer at the baseline and 12 weeks.
Change from baseline PE max (Maximal Expiratoy Pressure) (cm H2O) at 12 weeks | 12 weeks
  Change of PE max (Maximal Expiratoy Pressure) (cm H2O) will be measured on a computerized Spirometer at the baseline and 12 weeks.
Change from baseline FEV1/FVC % predicted at 12 weeks | 12 weeks
  Change of FEV1/FVC % Predicted (Percent Predicted of ratio of FEV1 and FVC) (% predicted) will be measured on a computerized Spirometer at the baseline and 12 weeks.
Change from baseline lower body strength assessed with Chair Standing test at 12 weeks | 12 weeks
  Change from baseline lower body strength assessed with Chair standing test. ( time/30 sec)
Change from baseline upper body strength assessed with Arm curl test at 12 weeks | 12 weeks
  Change from baseline upper body strength assessed with Arm curl test (time/30 sec)
Change from baseline lower body flexibility assessed with Chair Sit and Reach test at 12 weeks | 12 weeks
  Change from baseline lower body flexibility assessed with Chair Sit and Reach test (cm)
Change from baseline upper body flexibility assessed with Back Scratch test at 12 weeks | 12 weeks.
  Change from baseline upper body flexibility assessed with Back Scratch test (cm)
Change from baseline agility/dynamic balance assessed with 8-foot Up and Go test at 12 weeks | 12 weeks
  Change from baseline agility/dynamic balance assessed with 8-foot Up and Go test (sec)
Change from baseline Exercise Capacity assessed with 6-minute walk test at 12 weeks | 12 weeks
  Change from baseline Exercise Capacity assessed with 6-minute walk test (meter)

SECONDARY OUTCOMES:
Change from baseline Dyspnea score assessed with visual analog scale at 12 weeks | 12 weeks
  Dyspnea or shortness of breath will be measured by visual analog scale (VAS) 1-10 point scale at the baseline and 12 weeks.
Change from baseline Quality of life score assessed with St. George's respiratory Questionnaires (SGRQ) at 12 weeks. | 12 weeks
  Change from baseline Quality of Life score assessed with St. George's respiratory Questionnaires (SGRQ) in Thai version at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Amornpan Ajjimaporn, Ph.D, Study Chair — Mahidol
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No